CLINICAL TRIAL: NCT00677755
Title: Medical Termination of Pregnancy Due to Emergency Contraception Failure: A Randomized Trial Comparing Mifepristone Combined Misoprostol and Misoprostol Alone.
Brief Title: Medical Abortion for Emergency Contraception Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taizhou Hospital (Other)
Responsible Party: YiYang Zhu/Centra for Reproductive Medicine, Taizhou hospital of Zhejiang Province
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Taizhou2004-08
Record Dates: First submitted 2008-05-07; First posted 2008-05-14 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Emergency Contraception; Abortion, Induced
Keywords: Medical abortion; emergency contraception; mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mf+Ms (Experimental): The women in mifepristone combined misoprostol group (Mf+Ms) received a single dose of mifepristone (Mifepristone tablets; Xianju Pharmacy, Zhejiang, China) 200mg orally on day 1, and then returned to the clinic on day 3 and were given misoprostol (Cytotec tables; Searle,A Division of Monsanto.P.L.C, England )0.8mg orally
  Interventions: Drug: mifepristone combined misoprostol
- Ms-alone (Experimental): The control group (Ms-alone) patients were only administered 0.8 mg of misoprostol orally on day 3.
  Interventions: Drug: misoprostol alone protocol

INTERVENTIONS:
Drug: mifepristone combined misoprostol — women received a single dose of mifepristone (Mifepristone tablets; Xianju Pharmacy, Zhejiang, China) 200mg orally on day 1, and then returned to the clinic on day 3 and were given misoprostol (Cytotec tables; Searle,A Division of Monsanto.P.L.C, England )0.8mg orally
  Arms: Mf+Ms
Drug: misoprostol alone protocol — patients were only administered 0.8 mg of misoprostol orally on day 3.
  Arms: Ms-alone

SUMMARY:
The purpose of this study is to compare the efficacy, safety and acceptability of pre-treatment with mifepristone and misoprostol compared to misoprostol alone in the medical termination of pregnancy by mifepristone EC failure.

DETAILED DESCRIPTION:
Women usually request an abortion when they have experienced an emergency contraception (EC) failure; this population represents 13% of all early pregnancy terminations in China. Many women would prefer to choose a medical abortion in order to avoid anesthesia, over a surgical operation. However, medical termination of a pregnancy after mifepristone EC failure has not been studied although it has already been extensively practiced by empirical means in China. There is no clarification in literature as to whether mifepristone is still effective in medical abortion with its previous failure experience in EC. This randomized study was aimed to compare the efficacy, safety and acceptability of pre-treatment with mifepristone and misoprostol compared to misoprostol alone in the medical termination of pregnancy by mifepristone EC failure.

ELIGIBILITY:
Inclusion Criteria:

* Participants included in the study were women aged 16 years or older
* with good general health,
* experiencing a mifepristone emergency contraception failure,
* presenting an intrauterine singleton pregnancy confirmed by pelvic ultrasound scan, with a crown-rump length compatible within 56 days of gestation at the enrolled day, and
* seeking a medical abortion for unwanted pregnancy.
* Women who had a threatened abortion or a failure pregnancy were also included.
* Participants were required to sign an informed consent form before enrolment, willing to comply with the schedule of follow-up visits and willing to undergo surgical aspiration if indicated.

Exclusion Criteria:

* The exclusion criteria included suspected or proven ectopic pregnancy,
* allergy or contraindications for mifepristone (chronic systemic corticosteroid therapy, adrenal insufficiency) or misoprostol (hypertension, mitral stenosis, severe asthma, glaucoma, sickle cell anemia and hypotension),
* history or evidence of thromboembolism, cardiovascular disease or liver disease, hemoglobin ≤ 90 g/l, heavy smoking (more than 10 per day),
* presence of an intrauterine device, and breastfeeding.
* Other exclusion criteria included participants who had EC failure because incorrect use, for example, having further unprotected intercourse after EC.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 394 (Actual)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
complete abortion rate | study day 17 (14 days after misoprostol)

SECONDARY OUTCOMES:
side effects, timing of expulsion and duration of bleeding | timing of expulsion at day 17, others at 45day after abortion

CONTACTS AND LOCATIONS:
Overall Officials: YiYang Zhu, MD, Study Director — Centra for Reproductive Medicine of Taizhou hospital
Locations (1):
- Taizhou Hospital of zhejiang Province, Taizhou, Zhejiang, China